CLINICAL TRIAL: NCT01809392
Title: Decitabine Augments for Post Allogeneic Stem Cell Transplantation in Patients With Acute Myeloid Leukemia and Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hematology-02
Record Dates: First submitted 2013-01-18; First posted 2013-03-12 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Acute Myelocytic Leukemia; Myelodysplastic Syndromes
Keywords: Decitabine; hematopoietic stem cell transplant; Wilms' tumor 1; cytolytic T lymphocyte; Regulatory T cell
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Wilms Tumor | interventions — Decitabine

ARMS (2):
- decitabine (Experimental): 36 mg/m2 on day 42 after transplantation and administered daily for 5 consecutive days every 28 days for up to a total of 10 cycles
  Interventions: Drug: decitabine
- no decitabine (No Intervention)

INTERVENTIONS:
Drug: decitabine — 36 mg/m2 on day 42 after transplantation and administered daily for 5 consecutive days every 28 days for up to a total of 10 cycles
  Arms: decitabine

SUMMARY:
Allo - hematopoietic stem cell transplantation is currently the only way to cure myelodysplastic syndrome /acute leukemia . The existing experimental results showed that decitabine and 5-azacytidine up-regulated the expression of tumor Ags on leukemic blasts in vitro and expanded the numbers of immunomodulatory T regulatory cells in animal models. Reasoning that decitabine might selectively augment a graft versus leukemia effect, the investigators used decitabine administration after allogeneic stem cell transplantation to studied the immunologic sequelae.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed AML in complete or partial remission or MDS using WHO classification undergoing alloHSCT
* High resolution typing HLA-matched related or unrelated donor. Donors may be mismatched at single antigen at HLA-A, -B or -DR locus plus possible single antigen mismatch at HLA-C according to institution guidelines. Two-antigen mismatch at a single locus is not allowed.
* Age ≥ 18
* creatinine < 1.5 times the institutional ULN or creatinine clearance (calculated by the Cockroft and Gault method) ≥ 30 mL/min
* bilirubin < 1.5 times the institutional ULN
* AST, ALT and alkaline phosphatase < 2.5 times the institutional ULN.

Exclusion Criteria:

* History of previous alloHSCT prior to the current alloHSCT.
* Persistent AML or MDS after alloHSCT.
* Positive serology for HIV.
* Pregnancy or nursing.
* Other cancers less than or equal to 2 years prior study entry except: basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, prostate cancer stage T1a or T1b.
* Uncontrolled active infections requiring intravenous antibiotics. Clinically significant systemic illness (e.g. serious active infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), which, in the judgment of the Principal or Associate Investigator would compromise the patient's ability to tolerate protocol therapy.
* Known or suspected hypersensitivity to decitabine.
* Patients may not be receiving any other investigational agents.
* General or specific changes in patient's condition that render the patient unacceptable for further treatment in judgment of the investigators.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
To assess the effects of decitabine on graft versus leukemia post transplant. | three years

SECONDARY OUTCOMES:
To assess immunologic reconstitution after allo HSCT | three years

OTHER OUTCOMES:
To assess lymphoid and myeloid chimerism post transplantation | three years
To determine the incidence of acute and chronic GVHD | three years
To determine the rates disease relapse, 3-year disease-free survival, and overall survival | three years
To access the frequency of FoxP3+ CD4+CD25+ lymphocytes and WT1 specific CTL before and after decitabine treatment | three years
To assess changes in WT1 gene expression and methylation patterns before and after following decitabine treatment | three years

CONTACTS AND LOCATIONS:
Overall Officials: Fu chengcheng, Phd, Study Director — First Affiliated Hospital, Soochow University
Locations (1):
- First Affiliated Hospital, Soochow University, Suzhou, Jiangsu, China